CLINICAL TRIAL: NCT00377975
Title: Synergistic Induction of UCP-1 by Ephedrine/Caffeine and Pioglitazone: A Rationale for Combination Therapy of Obesity
Brief Title: "Pecos" B-adrenergic and PPAR-G Stimulation Upregulates Lipid Metabolism in Human Subcutaneous Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Steven Smith, Associate Professor, Adjunct, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 22021
Record Dates: First submitted 2006-09-17; First posted 2006-09-19 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: UCP-1; ephedrine; caffeine; pioglitazone
MeSH Terms: conditions — Obesity | interventions — Ephedrine; Pioglitazone; Caffeine

INTERVENTIONS:
Drug: Ephedrine
Drug: Pioglitazone
Drug: Caffeine

SUMMARY:
This study compares four treatments to see which one causes the most weight loss, fat loss, loss of abdominal fat and improvement in blood tests like cholesterol. The four treatments are: Placebo, Ephedrine plus caffeine, Pioglitazone, Combined pioglitazone and ephedrine plus caffeine

DETAILED DESCRIPTION:
The sympathetic nervous system, via the intracellular messenger cAMP and MAPK activation, and thiazolidinediones via PPARγ control lipid metabolism have been implicated in body weight regulation. The present study was undertaken to determine whether the simultaneous activation of these two signaling systems might synergize to exert beneficial effects on the expression of key genes involved in lipid metabolism and mitochondrial biogenesis in subcutaneous fat in healthy, non-diabetic subjects. Fifty seven non-diabetic women and men were randomized into four groups: 1) placebo/placebo (PP); 2) ephedrine plus caffeine/placebo (ECP); 3) placebo/pioglitazone (PPio); 4) ephedrine plus caffeine/pioglitazone (ECPio). Adipose tissue samples were obtained after 12 weeks of treatment to determine gene expression by real time RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* not pregnant or nursing
* using adequate contraception
* between 18 and 50 years of age
* BMI between 30 and 35 kg/m2

Exclusion Criteria:

* significant renal, cardiac, liver, lung or neurological disease
* high blood pressure
* diabetes
* prior use of thiazolidinedione
* prior use of beta-blockers alcohol or drug abuse
* history of thrombophlebitis, vascular or blood clotting disorders
* unwilling or unable to abstain from caffeinated beverages and alcohol prior to adipose tissue biopsy and metabolic rates measurements
* increased liver function test at baseline
* have metal objects that would interfere with the measurement of the body composition
* use drugs known to affect lipid metabolism, energy metabolism or body weight
* use herbal supplements containing ephedrine and/or caffeine
* take chronic medication, except hormone replacement or contraception
* are a woman unwilling to use effective contraception during the trial
* have heart disease or history of stroke
* have urinary symptoms from enlarged prostate
* have gained and or lost more than 10 pounds in the last 6 month
* have use a monoamine oxidase inhibitor medication in the last month
* have high or low thyroid function that has not been controlled in the normal range for at least 2 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96
Dates: Start 2003-01; Study Completion 2004-11

PRIMARY OUTCOMES:
Percent fat after 16 weeks treatment using a Hologic QDR 4500 DEXA.

SECONDARY OUTCOMES:
UCP-1 gene expression by quantitative RT-PCR
fat mass, lean mass
visceral adiposity by multi-slice CT scanning
resting metabolic rate and thermic effect of a single dose of ephedrine and caffeine
adipose tissue gene expression profiling using oligonucleotide array

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Pasarica M, Xie H, Hymel D, Bray G, Greenway F, Ravussin E, Smith SR. Lower total adipocyte number but no evidence for small adipocyte depletion in patients with type 2 diabetes. Diabetes Care. 2009 May;32(5):900-2. doi: 10.2337/dc08-2240. Epub 2009 Feb 19. PMID 19228873